CLINICAL TRIAL: NCT00065585
Title: Efficacy of Acupuncture for Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U01AT001110 (NIH); U01AT001110 (NIH)
Record Dates: First submitted 2003-07-28; First posted 2003-07-31 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Low Back Pain
Keywords: low back pain; acupuncture
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Usual care (No Intervention)
- non needle control (Placebo Comparator)
  Interventions: Procedure: Accupuncture
- Acupuncture - Standardized Points (Sham Comparator)
  Interventions: Procedure: Accupuncture
- Accupunture - Experimental Points (Experimental)
  Interventions: Procedure: Accupuncture

INTERVENTIONS:
Procedure: Accupuncture
  Arms: Accupunture - Experimental Points; Acupuncture - Standardized Points; non needle control

SUMMARY:
This is a trial to clarify the extent to which acupuncture needling can diminish the effect of chronic back pain on patient functioning and symptoms.

DETAILED DESCRIPTION:
This is a 4-arm multi-site randomized controlled trial to clarify the extent to which various types of acupuncture needling can diminish the effect of chronic low back pain on patient functioning and symptoms. Reviews have noted the poor quality of research in this area and urged that scientifically rigorous studies be conducted. Recent higher quality trials suggest acupuncture is a promising treatment for back pain. This study directly addresses methodological shortcomings that have plagued previous studies. A total of 640 subjects (160 per arm) with low back pain lasting at least 3 months will be recruited from group model HMOs in Seattle, WA and Oakland, CA. They will be randomized to one of three different methods of stimulation of acupuncture or to continue usual medical care. Ten treatments will be provided over 7 weeks. The primary outcomes, dysfunction and bothersomeness of low back pain, will be measured at baseline, and after 8, 26, and 52 weeks by telephone interviewers masked to treatment. Analysis of covariance within an intention-to-treat context will be used to analyze the data. Because chronic back pain is a major public health problem and the top reason patients seek acupuncture treatment, a clear, unambiguous assessment is critical for making informed decisions about whether acupuncture should be included as part of conventional care for back pain or covered by insurance. Results of this study will provide the clearest evidence to date about the value of acupuncture needling as a treatment for chronic low back pain.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of low back pain including lumbago, unspecified backache, sprains and strains of sacroiliac, lumbar, sacral, or unspecified regions of the spine
* Back pain must be of at least 3 months duration and rated at least 3 on a symptom bothersomeness scale

Exclusion criteria:

* non-mechanical causes or potential causes of low back pain (i.e. sciatica, underlying systemic or visceral disease, pregnancy, spondylolisthesis, spinal stenosis, cancer or unexplained weight loss, recent vertebral fracture)
* previous treatment with acupuncture
* inappropriate candidate for acupuncture (i.e. severe clotting disorders or on anticoagulant medication, heart pacemakers)
* characteristics complicating the interpretation of the findings (severe or progressive neurologic deficits, back surgery within the prior three years, planning to seek other treatment for back pain)
* characteristics related to ability to complete the study protocol (unable to speak English, plans to move out of town)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640
Dates: Start 2004-04; Primary Completion 2006-09 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cherkin, PhD, Study Director — Group Health Cooperative Center for Health Studies; Karen J Sherman, PhD, Principal Investigator — Group Health Cooperative Center for Health Studies; Andy Avins, MD, Principal Investigator — Kaiser Foundation Research Institute, Kaiser Permanente Northern California
Locations (2):
- United States (2):
  - Kaiser Permanente Northern California, Kaiser Foundation Research Institute, Oakland, California
  - Group Health Cooperative, Center for Health Studies, Seattle, Washington

REFERENCES:
- [Background] Cherkin DC, Sherman KJ, Hogeboom CJ, Erro JH, Barlow WE, Deyo RA, Avins AL. Efficacy of acupuncture for chronic low back pain: protocol for a randomized controlled trial. Trials. 2008 Feb 28;9:10. doi: 10.1186/1745-6215-9-10. PMID 18307808
- [Result] Cherkin DC, Sherman KJ, Avins AL, Erro JH, Ichikawa L, Barlow WE, Delaney K, Hawkes R, Hamilton L, Pressman A, Khalsa PS, Deyo RA. A randomized trial comparing acupuncture, simulated acupuncture, and usual care for chronic low back pain. Arch Intern Med. 2009 May 11;169(9):858-66. doi: 10.1001/archinternmed.2009.65. PMID 19433697
- [Derived] Sherman KJ, Hawkes RJ, Ichikawa L, Cherkin DC, Deyo RA, Avins AL, Khalsa PS. Comparing recruitment strategies in a study of acupuncture for chronic back pain. BMC Med Res Methodol. 2009 Oct 27;9:69. doi: 10.1186/1471-2288-9-69. PMID 19860906